CLINICAL TRIAL: NCT04732221
Title: A Phase 2/3, Multicenter, Randomized, Double-blind, Placebo-Controlled, Adaptive Design Study to Evaluate the Efficacy and Safety of MK-5475 in Adults With Pulmonary Arterial Hypertension
Brief Title: A Study of the Efficacy and Safety of Frespaciguat (MK-5475) in Participants With Pulmonary Arterial Hypertension (INSIGNIA-PAH: Phase 2/3 Study of an Inhaled sGC Stimulator in PAH) (MK-5475-007)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5475-007; MK-5475-007 (Other: MSD); 2022-500877-15-00 (Registry Identifier: EU CT); U1111-1278-4977 (Registry Identifier: UTN); 2020-001108-40 (EudraCT Number)
Record Dates: First submitted 2021-01-27; First posted 2021-02-01 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Arterial Hypertension; Hypertension, Pulmonary
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: A total of approximately 450 participants will be randomized in this operationally seamless adaptive Phase 2/3 study. Phase 2 of the study will randomize approximately 164 participants into 4 arms, and Phase 3 of the study will randomize approximately 286 participants into 2 arms.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 2 Cohort Frespaciguat 380 µg (Experimental): Participants receive frespaciguat 380 µg via oral inhalation once daily for 12 week base period and for optional 40 month extension period.
  Interventions: Drug: Frespaciguat
- Phase 2 Cohort Frespaciguat 100 µg (Experimental): Participants receive frespaciguat 100 µg via oral inhalation once daily for 12 week base period and for optional 40 month extension period.
  Interventions: Drug: Frespaciguat
- Phase 2 Cohort Frespaciguat 32 µg (Experimental): Participants receive frespaciguat 32 µg via oral inhalation once daily for 12 week base period and for optional 40 month extension period.
  Interventions: Drug: Frespaciguat
- Phase 2 Cohort Placebo (Placebo Comparator): Participants receive placebo via oral inhalation once daily for 12 week base period, and one of the MK-5475 doses (380, 100, or 32 µg) for the optional 40 month extension period.
  Interventions: Drug: Placebo to Frespaciguat
- Phase 3 Cohort Frespaciguat (Experimental): Participants receive one of 3 frespaciguat doses (380, 100 or 32 µg) to be selected at end of the Phase 2 Cohort, administered via oral inhalation once daily for 12-week base period and up to 40 months in the extension period
  Interventions: Drug: Frespaciguat
- Phase 3 Cohort Placebo (Placebo Comparator): Participants receive placebo via oral inhalation once daily for 12 week base period and up to 40 months in the extension period.
  Interventions: Drug: Placebo to Frespaciguat

INTERVENTIONS:
Drug: Frespaciguat — Frespaciguat (soluble guanylate cyclase stimulator) 380 µg, 100 µg or 32 µg administered as dry powder inhalation
  Arms: Phase 2 Cohort Frespaciguat 100 µg; Phase 2 Cohort Frespaciguat 32 µg; Phase 2 Cohort Frespaciguat 380 µg; Phase 3 Cohort Frespaciguat
Drug: Placebo to Frespaciguat — Placebo administered as dry powder inhalation
  Arms: Phase 2 Cohort Placebo; Phase 3 Cohort Placebo

SUMMARY:
This is a two-part (Phase 2/Phase 3) study of frespaciguat, an inhaled soluble guanylate cyclase stimulator, in participants with pulmonary arterial hypertension (PAH).

The first part (Phase 2) will assess three different doses of frespaciguat compared to placebo in a base period of 12 weeks, followed by comparison of three different doses of frespaciguat during an optional 40 month extension period. The treatment dose with the best efficacy and safety profile in the phase 2 cohort base period will be selected for use in the second part (Phase 3) of the study. The primary hypothesis of Phase 2 is that at least one frespaciguat dose is superior to placebo in reducing pulmonary vascular resistance (PVR) from baseline at week 12.

The purpose of the second part (Phase 3) of the study is to confirm the efficacy, safety, and tolerability of frespaciguat at the selected dose compared to placebo during a 12 week base period followed by an extension period of up to 5 years. The primary hypothesis of Phase 3 is that frespaciguat is superior to placebo in increasing 6-minute walk distance (6MWD) from baseline at week 12. Due to sponsor's decision this phase/part was not conducted.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary arterial hypertension (PAH) in one of the following groups:

  * Idiopathic PAH
  * Heritable PAH
  * Drug and toxin-induced PAH
  * PAH associated with connective tissue disease, HIV infection, or congenital heart disease.
* Diagnosis of PAH documented by right heart catheterization (RHC).
* Eligibility RHC meeting all of the following criteria:

  * Mean pulmonary artery pressure (mPAP) ≥25 mmHg
  * Pulmonary vascular resistance (PVR) of ≥3 Wood units
  * Pulmonary capillary wedge pressure (PCWP) or left ventricular end diastolic pressure (LVEDP) ≤15 mmHg.
* World Health Organization functional class (WHO-FC) symptoms between Class II and IV.
* Two 6-Minute walk distance (6MWD) measurements between 150 and 500 meters, one at screening and one at randomization.
* Stable concomitant background PAH-specific therapy.
* Body Mass Index (BMI) between 18.5 kg/m² and 40 kg/m² .
* Agree to be abstinent from heterosexual intercourse or use contraception during the intervention period and for at least 14 days after the last dose of study intervention.
* Female participants may not be pregnant or breastfeeding.

Exclusion Criteria:

* Group 2 to 5 pulmonary hypertension.
* PAH in one of the following groups:

  * Long term responders to calcium channel blockers
  * Overt features of venous/capillary involvement
* Evidence of more-than-mild obstructive lung disease.
* Evidence of more-than-mild parenchymal lung disease.
* Evidence of more-than-mild obstructive sleep apnea (OSA) that is untreated.
* Evidence or history of left heart disease, including any of the following:

  * Left ventricular ejection fraction (LVEF) ≤45%
  * Moderate or severe left-sided valvular disease (aortic or mitral valve stenosis or regurgitation)
  * Significant left ventricular diastolic dysfunction on echocardiographic evaluation
* Presence of 3 or more of the following risk factors for heart failure with preserved ejection fraction: BMI>30 kg/m², essential systemic hypertension, diabetes mellitus of any type, or coronary artery disease.
* Oxygen saturation measured by pulse oximetry (SpO₂) <90%, despite supplemental oxygen therapy.
* Chronic renal insufficiency (eGFR <30 mL/min)
* Chronic liver disease (i.e., Child-Pugh B or C), portal hypertension, cirrhosis, or significant hepatic laboratory abnormalities.
* Current smoker or currently uses electronic cigarettes (vapes).
* History of cancer, except: nonmelanomatous skin carcinoma or carcinoma in situ of the cervix or other malignancies which have been successfully treated, with appropriate follow up, and unlikely to recur for the duration of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (91):
- United States (26):
  - University of California San Diego Health-Pulmonary Critical Care ( Site 0061), La Jolla, California
  - University of California Davis Health-Internal Medicine: Pulmonary, Critical Care and Sleep Medicine, Sacramento, California
  - UCSF Helen Diller Medical Center at Parnassus Heights ( Site 0063), San Francisco, California
  - University of Colorado - Denver ( Site 0003), Aurora, Colorado
  - Cardiovascular Institute of North Colorado - Banner Health ( Site 0013), Greeley, Colorado
  - Georgetown University Hospital ( Site 0025), Washington D.C., District of Columbia
  - University of Miami Hospital-Division of Pulmonary & Critical Care ( Site 0053), Miami, Florida
  - AdventHealth Orlando ( Site 0040), Orlando, Florida
  - Tampa General Hospital ( Site 0058), Tampa, Florida
  - Indiana University Health Methodist Hospital ( Site 0045), Indianapolis, Indiana
  - University of Iowa Hospital and Clinics ( Site 0009), Iowa City, Iowa
  - University of Kansas Medical Center ( Site 0038), Kansas City, Kansas
  - University of Kentucky ( Site 0006), Lexington, Kentucky
  - Norton Pulmonary Specialists ( Site 0048), Louisville, Kentucky
  - University of Maryland ( Site 0032), Baltimore, Maryland
  - Washington University School of Medicine ( Site 0066), St Louis, Missouri
  - University of Nebraska Medical Center ( Site 0041), Omaha, Nebraska
  - University of New Mexico, Health Sciences Center ( Site 0028), Albuquerque, New Mexico
  - Clinical Trials Unit at Eastowne Medical Office Building ( Site 0019), Chapel Hill, North Carolina
  - AnMed Health ( Site 0033), Anderson, South Carolina
  - Statcare Pulmonary Consultants ( Site 0067), Knoxville, Tennessee
  - University of Texas Southwestern Medical Center at Dallas ( Site 0012), Dallas, Texas
  - Houston Methodist Research Institute ( Site 0036), Houston, Texas
  - The University of Texas Health Science Center at Houston ( Site 0054), Houston, Texas
  - Sentara Norfolk General Hospital ( Site 0014), Norfolk, Virginia
  - West Virginia University-WVU Heart and Vascular Institute ( Site 0051), Morgantown, West Virginia
- Argentina (8):
  - Cardiologia Palermo ( Site 0140), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Centro Medico Capital ( Site 0131), La Plata, Buenos Aires
  - Hospital Universitario Austral ( Site 0138), Pilar, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes ( Site 0141), Quilmes, Buenos Aires
  - Hospital El Cruce Nestor Carlos Kirchner ( Site 0132), San Juan Bautista, Buenos Aires
  - Sanatorio de la Trinidad Mitre ( Site 0130), Buenos Aires, Buenos Aires F.D.
  - Instituto Cardiovascular de Rosario ( Site 0128), Rosario, Santa Fe Province
  - Hospital Privado Universitario de Córdoba ( Site 0137), Córdoba
- Australia (3):
  - Nepean Hospital ( Site 0184), Kingswood, New South Wales
  - Macquarie University ( Site 0180), Macquarie University, New South Wales
  - John Hunter Hospital ( Site 0185), Newcastle, New South Wales
- Belgium (2):
  - Université Libre de Bruxelles - Hôpital Erasme ( Site 0601), Brussels, Bruxelles-Capitale, Region de
  - UZ Leuven ( Site 0600), Leuven, Vlaams-Brabant
- Canada (3):
  - Peter Lougheed Centre ( Site 0107), Calgary, Alberta
  - University Health Network - Toronto General Hospital ( Site 0104), Toronto, Ontario
  - IUCPQ ( Site 0111), Québec, Quebec
- Colombia (3):
  - Centro Cardiovascular Colombiano Clínica Santa María ( Site 0154), Medellín, Antioquia
  - Hospital Universitario San Ignacio ( Site 0152), Bogotá, Bogota D.C.
  - Fundacion Cardiovascular de Colombia ( Site 0155), Piedecuesta, Santander Department
- France (5):
  - CHRU Brest - Hopital Cavale Blanche ( Site 0254), Brest, Finistere
  - CHU de Toulouse - Hopital Larrey ( Site 0258), Toulouse, Haute-Garonne
  - Institut Coeur Poumon - CHRU de Lille ( Site 0252), Lille, Hauts-de-France
  - Centre Hospitalier Universitaire de Rouen ( Site 0253), Rouen, Seine-Maritime
  - CHU - Hopital de Bicetre ( Site 0251), Le Kremlin-Bicêtre, Val-de-Marne
- Germany (6):
  - Thoraxklinik Heidelberg gGmbH am Universitaetsklinikum Heidelberg ( Site 0276), Heidelberg, Baden-Wurttemberg
  - Klinikum Würzburg Mitte-Medizinische Klinik - Schwerpunkt Pneumologie & Beatmungsmedizin ( Site 0280, Würzburg, Bavaria
  - UKGM Gießen/Marburg ( Site 0279), Giessen, Hesse
  - Medizinische Hochschule Hannover ( Site 0284), Hanover, Lower Saxony
  - Uniklinikum Dresden ( Site 0283), Dresden, Saxony
  - Universitaetsklinikum Leipzig ( Site 0285), Leipzig, Saxony
- AHEPA University General Hospital of Thessaloniki ( Site 0577), Thessaloniki, Greece
- Israel (5):
  - Soroka Medical Center ( Site 0330), Beersheba
  - Rambam Medical Center ( Site 0335), Haifa
  - Wolfson Medical Center [Holon, Israel] ( Site 0333), Holon
  - Shaare Zedek Medical Center ( Site 0331), Jerusalem
  - Rabin Medical Center ( Site 0327), Petah Tikva
- Italy (5):
  - University of Naples Federico II ( Site 0308), Naples, Campania
  - Azienda Ospedaliera Policlinico Umberto I ( Site 0301), Rome, Lazio
  - Ospedale San Gerardo - ASST Monza ( Site 0304), Monza, Monza E Brianza
  - Centro Cardiologico Monzino IRCCS ( Site 0306), Milan
  - Fondazione IRCCS Policlinico San Matteo ( Site 0302), Pavia
- Mexico (3):
  - Instituto Nacional de Cardiología -Ignacio Chavez ( Site 0651), Mexico City, Mexico City
  - Consultorio 1020 Hospital Angeles Xalapa ( Site 0654), Xalapa, Veracruz
  - Operadora de Hospitales Angeles. S.A. de C.V. -Sucursal Lomas ( Site 0653), Huixquilucan
- New Zealand (2):
  - Christchurch Hospital ( Site 0201), Christchurch, Canterbury
  - Greenlane Clinical Centre ( Site 0203), Auckland
- Poland (3):
  - Krakowski Szpital Specjalistyczny im. Jana Pawa II-Oddzial Kliniczny Chorob Serca i Naczyn z Pododd, Krakow, Lesser Poland Voivodeship
  - Specjalistyczny Szpital im. Dr Alfreda Sokolowskiego w Walbrzychu ( Site 0351), Wałbrzych, Lower Silesian Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie ( Site 0352), Lublin, Lublin Voivodeship
- Russia (2):
  - Scientific Research Institute Complex Problems Cardiovascular Disease ( Site 0403), Kemerovo, Kemerovo Oblast
  - Almazov National Medical Research Centre of the Ministry of Health ( Site 0402), Saint Petersburg, Sankt-Peterburg
- Sweden (2):
  - Akademiska sjukhuset ( Site 0453), Uppsala, Uppsala County
  - Sahlgrenska Universitetssjukhuset-Cardiology Research Unit ( Site 0452), Gothenburg, Västra Götaland County
- Turkey (Türkiye) (8):
  - Ege Universitesi Hastanesi-Cardilogy Department ( Site 0504), Bornova, İzmir
  - Hacettepe Universitesi Tip Fakultesi Hastanesi ( Site 0510), Ankara
  - Akdeniz Uni.Tip Fakultesi Saglik Uygulama ve Arastirma Merkezi ( Site 0508), Antalya
  - Eskisehir Osmangazi Uni. Tip Fakultesi Hastanesi ( Site 0506), Eskişehir
  - Istanbul Uni. Kardiyoloji Enstitusu ( Site 0502), Istanbul
  - Istanbul Universitesi Istanbul Tip Fakultesi ( Site 0509), Istanbul
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi ( Site 0501), Istanbul
  - Dokuz Eylul University Faculty of Medicine ( Site 0505), Izmir
- United Kingdom (4):
  - Golden Jubilee National Hospital ( Site 0556), Glasgow, Glasgow City
  - Royal Brompton and Harefield NHS Trust ( Site 0553), London, London, City of
  - Imperial College Healthcare NHS Trust - Hammersmith Hospital ( Site 0554), London, London, City of
  - The Freeman Hosp.Newcastle upon Tyne Hosp NHS Trust ( Site 0552), Newcastle upon Tyne, Newcastle Upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Humbert M, Hassoun PM, Chin KM, Bortman G, Patel MJ, La Rosa C, Fu W, Loureiro MJ, Hoeper MM. MK-5475, an inhaled soluble guanylate cyclase stimulator, for treatment of pulmonary arterial hypertension: the INSIGNIA-PAH study. Eur Respir J. 2024 Nov 14;64(5):2401110. doi: 10.1183/13993003.01110-2024. Print 2024 Nov. PMID 39255991
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26191&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was planned to be conducted in 2 parts: a Phase 2 dose selection cohort and a Phase 3 confirmatory cohort. Due to sponsor's decision, Phase 3 was not conducted.
Groups:
- Base Period: Placebo: Participants received placebo via oral inhalation once daily for 12 week base period
- Base Period: MK-5475 32 µg: Participants received MK-5475 32 µg via oral inhalation once daily for 12 week base period
- Base Period: MK-5475 100 µg: Participants received MK-5475 100 µg via oral inhalation once daily for 12 week base period
- Base Period: MK-5475 380 µg: Participants receive MK-5475 380 µg via oral inhalation once daily for 12 week base period
- Extension Period: MK-5475 32 µg: Participants who received MK-3475 32 ug in the base period, and participants who received placebo in the base period and were randomized to the 32 ug group in the extension period, were administered MK-3475 32ug via oral inhalation for up to 25 months
- Extension Period: MK-5475 100 µg: Participants who received MK-3475 100 ug in the base period, and participants who received placebo in the base period and were randomized to the 100 ug group in the extension period, were administered MK-3475 100 ug via oral inhalation for up to 25 months
- Extension Period: MK-5475 380 μg: Participants who received MK-3475 380 ug in the base period, and participants who received placebo in the base period and were randomized to the 380 ug group in the extension period, were administered MK-3475 380 ug via oral inhalation for up to 25 months
Period: Base Period
Arm/Group | Base Period: Placebo | Base Period: MK-5475 32 µg | Base Period: MK-5475 100 µg | Base Period: MK-5475 380 µg | Extension Period: MK-5475 32 µg | Extension Period: MK-5475 100 µg | Extension Period: MK-5475 380 μg
Started | 41 | 42 | 44 | 41 | 0 | 0 | 0
Completed | 39 | 41 | 43 | 41 | 0 | 0 | 0
Not Completed | 2 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 0 | 0
Period: Extension Period
Arm/Group | Base Period: Placebo | Base Period: MK-5475 32 µg | Base Period: MK-5475 100 µg | Base Period: MK-5475 380 µg | Extension Period: MK-5475 32 µg | Extension Period: MK-5475 100 µg | Extension Period: MK-5475 380 μg
Started | 0 | 0 | 0 | 0 | 45 | 46 | 44
Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 44 | 46 | 44
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Sponsors Decision | 0 | 0 | 0 | 0 | 41 | 40 | 40
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Base Period: Placebo | Base Period: MK-5475 32 µg | Base Period: MK-5475 100 µg | Base Period: MK-5475 380 µg | Total
Number analyzed (Participants) | 41 | 42 | 44 | 41 | 168
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.1 (12.7) | 48.1 (16.9) | 51.7 (14.2) | 47.6 (15.9) | 49.9 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 34 | 32 | 30 | 124
  Male | 13 | 8 | 12 | 11 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 14 | 10 | 12 | 47
  Not Hispanic or Latino | 30 | 27 | 33 | 29 | 119
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 0 | 0 | 3
  Asian | 3 | 1 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 1 | 1 | 7
  White | 32 | 34 | 41 | 36 | 143
  More than one race | 1 | 4 | 2 | 4 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 2 Cohort: Mean Percent Change From Baseline in Pulmonary Vascular Resistance (PVR) at 12 Weeks
Description: PVR was calculated in participants after MK-5475 dosing at baseline and Week 12. PVR is assessed by right heart catheterization (RHC). Based on the variables obtained by right heart catheterization (RHC), the percentage change from baseline PVR was calculated. Per protocol, this outcome measure was assessed only for base period and was not assessed during extension period.
Time Frame: At baseline and 12 weeks
Population: All randomized participants who received ≥1 dose of study treatment and had baseline observation.
Measure: Least Squares Mean (Standard Error); unit: Percentage Change
Arm/Group | Base Period: Placebo | Base Period: MK-5475 32 µg | Base Period: MK-5475 100 µg | Base Period: MK-5475 380 µg
Number analyzed (Participants) | 41 | 42 | 44 | 41
Percentage Change | 4.3 (4.45) | -4.9 (4.07) | -17.6 (4.07) | -15.6 (5.39)
Statistical Analysis 1: Comparison: Base Period: Placebo vs Base Period: MK-5475 32 µg; Test type: Superiority; p = 0.068, Robust Regression — A 1-sided p-value was obtained from fitting a Robust regression estimate based on a Huber-type M estimator including terms for treatment and WHO-FC (Class II and Class III/IV) at baseline; Missing data at week 12 due to death were imputed using the worst observed value and other missingness were imputed using J2R method; Treatment difference = -9.2, 95% CI 2-sided [-21.3 to 2.9] — Least Square Mean of the overall treatment difference with 95% confidence interval (CI) was reported
Statistical Analysis 2: Comparison: Base Period: Placebo vs Base Period: MK-5475 100 µg; Test type: Superiority; p < 0.001, Robust Regression — based on a Huber-type M estimator including terms for treatment and WHO-FC (Class II and Class III/IV) at baseline; [statistical method as in outcome 1, analysis 1]; Treatment difference = -22.0, 95% CI 2-sided [-33.7 to -10.3] — Least Square Mean of the overall treatment difference with 95% confidence interval (CI) was reported
Statistical Analysis 3: Comparison: Base Period: Placebo vs Base Period: MK-5475 380 µg; Test type: Superiority; p = 0.002, Robust Regression — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Treatment difference = -19.9, 95% CI 2-sided [-33.4 to -6.4] — Least Square Mean of the overall treatment difference with 95% confidence interval (CI) was reported

2. Primary Outcome: Phase 3 Cohort: Mean Change From Baseline in 6-Minute Walk Distance (6MWD) at 12 Weeks
Description: 6MWD is measured by an exercise test known as 6-Minute Walk Test (6MWT) that assesses functional capacity. It measures the distance covered over a time of 6 minutes and is intended to be used as an outcome measure by which to compare changes in excercise capacity. Each participant's 6MWD is to be measured at baseline and at 12 weeks. An increase in the distance walked during the 6MWT indicates improvement in functional exercise capacity.
Time Frame: At baseline and 12 weeks
Population: Phase 3 was not conducted due to the sponsor's decision and thus no data were collected for the outcome measure.
Groups:
- Extension Period: MK-5475 32 µg: Participants who received MK-5475 32 μg in the base period, and those who received matching placebo for MK-5475 32 μg at the end of the base period (12 weeks) were administered MK-5475 32 μg via oral inhalation up to 25 months in the extension period
Arm/Group | Base Period: Placebo | Base Period: MK-5475 32 µg | Base Period: MK-5475 100 µg | Base Period: MK-5475 380 µg | Extension Period: MK-5475 32 µg | Extension Period: MK-5475 100 µg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Phase 2 Cohort: Mean Change From Baseline in 6-Minute Walk Distance (6MWD) at 12 Weeks
Description: 6MWD is measured by an exercise test known as 6-Minute Walk Test (6MWT) that assesses functional capacity. It measures the distance covered over a time of 6 minutes and is used as an outcome measure by which to compare changes in exercise capacity. Each participant's 6MWD was measured at baseline and at 12 weeks. An increase in the distance walked during the 6MWT indicates improvement in functional exercise capacity.
Time Frame: At baseline and 12 weeks
Population: All randomized participants in Phase 2 who received ≥1 dose of study treatment and had baseline observation.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Base Period: Placebo | Base Period: MK-5475 32 µg | Base Period: MK-5475 100 µg | Base Period: MK-5475 380 µg
Number analyzed (Participants) | 38 | 41 | 42 | 40
Meters | 24.6 (66.3) | 27.4 (53.1) | 10.8 (45.6) | 11.3 (38.9)

4. Secondary Outcome: Phase 2 Cohort: Mean Change From Baseline in Mean Right Atrial Pressure (mRAP) at 12 Weeks
Description: mRAP is the blood pressure in the right atrium of the heart. mRAP was assessed by right heart catheterization (RHC).A decrease in mRAP indicates improvement in right ventricular function, reduction of PAH related morbidity.
Time Frame: At baseline and 12 weeks
Population: All randomized participants in Phase 2 who received ≥1 dose of study treatment and had baseline observation.
Measure: Mean (Full Range); unit: Millimeters of Mercury (mmHg)
Arm/Group | Base Period: Placebo | Base Period: MK-5475 32 µg | Base Period: MK-5475 100 µg | Base Period: MK-5475 380 µg
Number analyzed (Participants) | 36 | 41 | 41 | 40
Millimeters of Mercury (mmHg) | 0.3 [-8.0 to 9.0] | 0.3 [-17.0 to 7.0] | -0.5 [-8.0 to 14.0] | -0.1 [-14.0 to 12.0]

5. Secondary Outcome: Phase 2 Cohort: Mean Change From Baseline in Cardiac Index (CI) at 12 Weeks
Description: The cardiac index (CI) is a hemodynamic measure that represents the cardiac output (CO) of an individual divided by their body surface area (BSA). Cardiac index is assessed by right heart catheterization (RHC). An increase in CI is indicates better right ventricular function and is associated with a reduction of PAH related morbidity and mortality.
Time Frame: At baseline and 12 weeks
Population: All randomized participants in Phase 2 who received ≥1 dose of study treatment and had baseline observation.
Measure: Mean (Full Range); unit: Liter/minutes/meter square (L/min/m^2)
Arm/Group | Base Period: Placebo | Base Period: MK-5475 32 µg | Base Period: MK-5475 100 µg | Base Period: MK-5475 380 µg
Number analyzed (Participants) | 37 | 40 | 41 | 41
Liter/minutes/meter square (L/min/m^2) | 0.1 [-0.9 to 3.1] | 0.0 [-1.7 to 1.4] | 0.2 [-1.4 to 1.5] | 0.1 [-1.6 to 1.8]

6. Secondary Outcome: Phase 2 Cohort: Mean Change From Baseline in Stroke Volume Index (SVI) at 12 Weeks
Description: The stroke volume index represents the amount of blood in mL, per square meter of body surface area, that is mobilized with each heart beat. SVI is assessed by RHC. An increase in SVI indicates better right ventricular function and is associated with a reduction of PAH related morbidity and mortality.
Time Frame: At baseline and 12 weeks
Population: All randomized participants in Phase 2 who received ≥1 dose of study treatment and had baseline observation.
Measure: Mean (Full Range); unit: mL/beat/m^2
Arm/Group | Base Period: Placebo | Base Period: MK-5475 32 µg | Base Period: MK-5475 100 µg | Base Period: MK-5475 380 µg
Number analyzed (Participants) | 37 | 40 | 41 | 41
mL/beat/m^2 | 2.9 [-9.3 to 44.4] | 0.2 [-37.2 to 20.7] | 3.2 [-21.8 to 35.2] | 1.2 [-29.1 to 25.1]

7. Secondary Outcome: Phase 3 Cohort: Mean Change From Baseline in 6-Minute Walk Distance (6MWD) at 24 Weeks
Description: 6MWD is measured by an exercise test known as 6-Minute Walk Test (6MWT) that assesses functional capacity. It measures the distance covered over a time of 6 minutes and is intended to be used as an outcome measure by which to compare changes in exercise capacity. Each participant's 6MWD is to be measured at baseline and at 24 weeks. An increase in the distance walked during the 6MWT indicates improvement in functional exercise capacity.
Time Frame: At baseline and 24 weeks
Population: Phase 3 was not conducted due to the sponsor's decision and thus no data were collected for the outcome measure.
Arm/Group | Base Period: Placebo | Base Period: MK-5475 32 µg | Base Period: MK-5475 100 µg | Base Period: MK-5475 380 µg | Extension Period: MK-5475 32 µg | Extension Period: MK-5475 100 µg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Phase 3 Cohort: Proportion of Participants Whose World Health Organization Functional Class (WHO-FC) is Not Worse at 12 Week Relative to Baseline
Description: The World Health Organization (WHO) classification of functional status is a measure of disease severity, based on a patient's description of their level of functioning and symptoms of disease in relation to their everyday activity. Patients were to be assigned 1 of 4 WHO-FC, dependent on limits of physical activity. As WHO-FC increases from I to IV, limits of physical activity were to increase.
Time Frame: At baseline and 12 weeks
Population: Phase 3 was not conducted due to the sponsor's decision and thus no data were collected for the outcome measure.
Arm/Group | Base Period: Placebo | Base Period: MK-5475 100 µg | Base Period: MK-5475 32 µg | Base Period: MK-5475 380 µg | Extension Period: MK-5475 32 µg | Extension Period: MK-5475 100 µg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Phase 2 Cohort: Number of Participants Who Experienced an Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Time Frame: Up to approximately 2.25 years
Population: Analysis population consisted of all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Base Period: Placebo | Base Period: MK-5475 32 µg | Base Period: MK-5475 100 µg | Base Period: MK-5475 380 µg | Extension Period: MK-5475 32 µg | Extension Period: MK-5475 100 µg | Extension Period: MK-5475 380 μg
Number analyzed (Participants) | 41 | 42 | 44 | 41 | 45 | 44 | 44
Participants | 27 | 28 | 28 | 27 | 33 | 38 | 39

10. Secondary Outcome: Phase 2 Cohort: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued treatment due to an AE was assessed.
Time Frame: Up to approximately 2.25 years
Population: Analysis population consisted of all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Base Period: Placebo | Base Period: MK-5475 32 µg | Base Period: MK-5475 100 µg | Base Period: MK-5475 380 µg | Extension Period: MK-5475 32 µg | Extension Period: MK-5475 100 µg | Extension Period: MK-5475 380 μg
Number analyzed (Participants) | 41 | 42 | 44 | 41 | 45 | 44 | 44
Participants | 0 | 1 | 0 | 0 | 0 | 1 | 0

11. Secondary Outcome: Phase 3 Cohort: Number of Participants Who Experienced an Adverse Event
Description: as for outcome 9
Time Frame: Up to approximately 2.25 years
Population: Phase 3 was not conducted due to the sponsor's decision and thus no data were collected for the outcome measure.
Arm/Group | Base Period: Placebo | Base Period: MK-5475 32 µg | Base Period: MK-5475 100 µg | Base Period: MK-5475 380 µg | Extension Period: MK-5475 32 µg | Extension Period: MK-5475 100 µg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Phase 3 Cohort: Number of Participants Who Discontinued Study Drug Due to an AE
Description: as for outcome 10
Time Frame: Up to approximately 2.25 years
Population: Phase 3 was not conducted due to the sponsor's decision and thus no data were collected for the outcome measure.
Arm/Group | Base Period: Placebo | Base Period: MK-5475 32 µg | Base Period: MK-5475 100 µg | Base Period: MK-5475 380 µg | Extension Period: MK-5475 32 µg | Extension Period: MK-5475 100 µg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 37 months
Description: All-cause mortality includes all randomized participants and adverse events include all participants who received at least one dose of study treatment.
Groups:
- Base Period: MK-5475 380 µg: Participants received MK-5475 380 µg via oral inhalation once daily for 12 week base period
- Extension Period: Placebo to MK-5475 32 µg: Participants who received placebo for the during the 12 week base period and were randomized to MK-3475 32 ug for the extension period, received MK-3475 32 ug via oral inhalation once daily for up to 25 months
- Extension Period: Placebo to MK-5475 100 µg: Participants who received placebo for the during the 12 week base period and were randomized to MK-3475 100 ug for the extension period, received MK-3475 100 ug via oral inhalation once daily for up to 25 months
- Extension Period: Placebo to MK-5475 380 µg: Participants who received placebo for the during the 12 week base period and were randomized to MK-3475 380 ug for the extension period, received MK-3475 380 ug via oral inhalation once daily for up to 25 months
- Extension Period: MK-5475 32 µg: Participants who received MK-3475 32 ug during the 12 week base period, received MK-3475 32 ug via oral inhalation once daily for up to 25 months
- Extension Period: MK-5475 100 µg: Participants who received MK-3475 100 ug during the 12 week base period, received MK-3475 100 ug via oral inhalation once daily for up to 25 months
- Extension Period: MK-5475 380 μg: Participants who received MK-3475 380 ug during the 12 week base period, received MK-3475 380 ug via oral inhalation once daily for up to 25 months
Arm/Group | Base Period: Placebo | Base Period: MK-5475 32 µg | Base Period: MK-5475 100 µg | Base Period: MK-5475 380 µg | Extension Period: Placebo to MK-5475 32 µg | Extension Period: Placebo to MK-5475 100 µg | Extension Period: Placebo to MK-5475 380 µg | Extension Period: MK-5475 32 µg | Extension Period: MK-5475 100 µg | Extension Period: MK-5475 380 μg
All-Cause Mortality (participants affected / at risk) | 2/41 | 0/42 | 1/44 | 0/41 | 1/11 | 0/9 | 0/10 | 0/34 | 0/37 | 2/34
Serious Adverse Events (participants affected / at risk) | 5/41 | 4/42 | 3/44 | 4/41 | 3/11 | 2/9 | 4/10 | 5/34 | 4/37 | 11/34
Other Adverse Events (participants affected / at risk) | 18/41 | 22/42 | 23/44 | 21/41 | 7/11 | 7/9 | 8/10 | 24/34 | 28/37 | 28/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Base Period: Placebo (N=41) | Base Period: MK-5475 32 µg (N=42) | Base Period: MK-5475 100 µg (N=44) | Base Period: MK-5475 380 µg (N=41) | Extension Period: Placebo to MK-5475 32 µg (N=11) | Extension Period: Placebo to MK-5475 100 µg (N=9) | Extension Period: Placebo to MK-5475 380 µg (N=10) | Extension Period: MK-5475 32 µg (N=34) | Extension Period: MK-5475 100 µg (N=37) | Extension Period: MK-5475 380 μg (N=34)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular device occlusion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Device leakage (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aneurysm thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Base Period: Placebo (N=41) | Base Period: MK-5475 32 µg (N=42) | Base Period: MK-5475 100 µg (N=44) | Base Period: MK-5475 380 µg (N=41) | Extension Period: Placebo to MK-5475 32 µg (N=11) | Extension Period: Placebo to MK-5475 100 µg (N=9) | Extension Period: Placebo to MK-5475 380 µg (N=10) | Extension Period: MK-5475 32 µg (N=34) | Extension Period: MK-5475 100 µg (N=37) | Extension Period: MK-5475 380 μg (N=34)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blindness unilateral (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 3 (4) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 1 (1) | 2 (3)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 2 (3) | 3 (4) | 1 (1)
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 2 (3)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (6)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial disease carrier (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 5 (5) | 6 (6) | 6 (7)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 5 (5) | 2 (2)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 4 (5) | 4 (6) | 4 (4)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 3 (3)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 3 (8) | 2 (2) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 8 (10) | 2 (2) | 3 (8)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (6) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 3 (10) | 2 (2) | 2 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 5 (6) | 4 (5) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 3 (3) | 8 (8) | 6 (7) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 8 (8) | 4 (6)
Product after taste (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 4 (5) | 4 (4) | 5 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 6 (7) | 2 (3) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 3 (3) | 1 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (3) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 3 (3)
Venous occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT04732221/Prot_SAP_000.pdf